CLINICAL TRIAL: NCT02396017
Title: Split-dose Versus Single-dose Polyethylene Glycol Regimen for Capsule Endoscopy Is Timing of Preparation for Capsule Endoscopy the Key for the Best Small-bowel Cleansing?
Brief Title: Split-dose Versus Single-dose Polyethylene Glycol Regimen for Capsule Endoscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Hospitalar Lisboa Ocidental (Other Government)
Responsible Party: Principal Investigator, Pedro Magalhães-Costa, MD, Centro Hospitalar Lisboa Ocidental
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SPLIT-PEG-CE
Record Dates: First submitted 2015-02-18; First posted 2015-03-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Bowel Preparation
MeSH Terms: interventions — Capsule Endoscopy; Polyethylene Glycols

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single-dose Polyethylene Glycol regimen (Active Comparator): Drug: Polyethylene Glycol Intervention: 2 liters of Polyethylene Glycol will be given in the day before Capsule Endoscopy ingestion.
  Interventions: Device: Capsule endoscopy; Drug: Polyethylene Glycol
- Split-dose Polyethylene Glycol regimen (Experimental): Drug: Polyethylene Glycol Intervention: 1 liter of Polyethylene Glycol will be given in the day before Capsule Endoscopy ingestion and another 1 liter Polyethylene Glycol will be given in the same day of Capsule Endoscopy ingestion.
  Interventions: Device: Capsule endoscopy; Drug: Polyethylene Glycol

INTERVENTIONS:
Device: Capsule endoscopy — Endoscopic device
Drug: Polyethylene Glycol — Bowel purgative
  Other Names: PEG

SUMMARY:
To compare the small bowel cleanliness for wireless capsule endoscopy using two different Polyethylene Glycol administration schedules (before the wireless capsule endoscopy ingestion versus in a split-dose fashion).

DETAILED DESCRIPTION:
The image quality obtained from the wireless capsule endoscopy improves its diagnostic yield. The amount of visualized mucosa is in direct correlation with the diagnostic yield. Nonetheless, frequently, the quality of the image obtained is hampered by the presence of bubbles, debris, bile and enteric fluid. Therefore many efforts have been putted in order to eliminate this factor such as the use of prokinetics, simethicone and bowel purgatives. The latter (namely the polyethylene glycol - PEG - solution) has accumulated evidence and is, therefore, recommended by the last European guidelines. Usually, the cleansing starts and finish in the day before the capsule endoscopy ingestion.

We hypothesized that, similarly to what had become evidence to large bowel cleansing, a shorter gap between the polyethylene glycol intake and the exam could provide a better capsule endoscopy image quality and therefore gauging our diagnostic yield.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients referred to our institution for CE during the study period

Exclusion Criteria:

* inpatients, bedridden, patients with clinical evidence of active bleeding, past history of abdominal surgery, abdominal or pelvic radiation therapy, occlusion, bowel perforation (suspected or confirmed), use of oral iron replacement therapy, severe cardiopulmonary, renal or hepatic disease, pregnancy, hypersensitivity to any components of the preparation, patients that didn't complete the preparation protocol, patients with incomplete enteroscopies (a complete enteroscopy is defined by the visualization of the mucosa from the duodenal bulb to the cecum), patients enrolled in other clinical studies and patients who didn't signed informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Small-bowel cleanliness | at the end of capsule endoscopy exploration
  The cleansing quality of the small-bowel will be evaluated according to the system validated by Brotz et al., using the quantitative index (QI), because this score is less susceptible to the subjective element. The used cut-off value accepted for an adequate small-bowel cleansing was ≥ 8 points.

SECONDARY OUTCOMES:
The number of all the observed lesions | at the end of capsule endoscopy exploration
  Estimate the number of all the observed lesions on the recording according to their hemorrhagic potential.
The clinical tolerance questionnaire | at the end of capsule endoscopy exploration
  Evaluate the clinical tolerance and the acceptability of the bowel preparation with the oral polyethylene glycol solution.
The transit time | at the end of capsule endoscopy exploration
  Compare gastric transit time and the small bowel transit time.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Chagas, MD, Study Director — Gastroenterology Department, Hospital Egas Moniz, Centro Hospitalar Lisboa Ocidental
Locations (1):
- Gastroenterology Department, Hospital Egas Moniz, Lisbon, Lisbon District, Portugal

REFERENCES:
- [Background] Rokkas T, Papaxoinis K, Triantafyllou K, Pistiolas D, Ladas SD. Does purgative preparation influence the diagnostic yield of small bowel video capsule endoscopy?: A meta-analysis. Am J Gastroenterol. 2009 Jan;104(1):219-27. doi: 10.1038/ajg.2008.63. PMID 19098872
- [Background] Ladas SD, Triantafyllou K, Spada C, Riccioni ME, Rey JF, Niv Y, Delvaux M, de Franchis R, Costamagna G; ESGE Clinical Guidelines Committee. European Society of Gastrointestinal Endoscopy (ESGE): recommendations (2009) on clinical use of video capsule endoscopy to investigate small-bowel, esophageal and colonic diseases. Endoscopy. 2010 Mar;42(3):220-7. doi: 10.1055/s-0029-1243968. Epub 2010 Mar 1. PMID 20195992
- [Background] Brotz C, Nandi N, Conn M, Daskalakis C, DiMarino M, Infantolino A, Katz LC, Schroeder T, Kastenberg D. A validation study of 3 grading systems to evaluate small-bowel cleansing for wireless capsule endoscopy: a quantitative index, a qualitative evaluation, and an overall adequacy assessment. Gastrointest Endosc. 2009 Feb;69(2):262-70, 270.e1. doi: 10.1016/j.gie.2008.04.016. Epub 2008 Oct 11. PMID 18851851
- [Background] Hassan C, Bretthauer M, Kaminski MF, Polkowski M, Rembacken B, Saunders B, Benamouzig R, Holme O, Green S, Kuiper T, Marmo R, Omar M, Petruzziello L, Spada C, Zullo A, Dumonceau JM; European Society of Gastrointestinal Endoscopy. Bowel preparation for colonoscopy: European Society of Gastrointestinal Endoscopy (ESGE) guideline. Endoscopy. 2013;45(2):142-50. doi: 10.1055/s-0032-1326186. Epub 2013 Jan 18. PMID 23335011
- [Derived] Magalhaes-Costa P, Carmo J, Bispo M, Santos S, Chagas C. Superiority of the Split-dose PEG Regimen for Small-Bowel Capsule Endoscopy: A Randomized Controlled Trial. J Clin Gastroenterol. 2016 Aug;50(7):e65-70. doi: 10.1097/MCG.0000000000000460. PMID 26646803